CLINICAL TRIAL: NCT03894449
Title: Probing the Synergistic Effect of Pre-Biotics & Iron Fortificants in Anemic
Brief Title: Probing the Synergistic Effect of Pre-Biotics & Iron Fortificants in Anemic Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, ABDUL MOMIN RIZWAN AHMAD, Principal Investigator, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-VA-04
Record Dates: First submitted 2019-03-25; First posted 2019-03-28 (Actual); Results first posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo only (Placebo Comparator)
  Interventions: Combination Product: Prebiotic + Iron Forificant
- Prebiotic Inulin & Iron Salt FeSO4 (Experimental)
  Interventions: Combination Product: Prebiotic + Iron Forificant
- Prebiotic GOS & Iron Salt FeSO4 (Experimental)
  Interventions: Combination Product: Prebiotic + Iron Forificant
- Prebiotic Inulin & Iron Salt NaFeEDTA (Experimental)
  Interventions: Combination Product: Prebiotic + Iron Forificant
- Prebiotic GOS & Iron Salt NaFeEDTA (Experimental)
  Interventions: Combination Product: Prebiotic + Iron Forificant

INTERVENTIONS:
Combination Product: Prebiotic + Iron Forificant — A combination dosage of prebiotic (Inulin or GOS) and Iron Fortificant (FeSO4 or NaFeEDTA) will be given to the study subjects.

SUMMARY:
Hypothesis: Synergistic effect of pre-biotics and iron fortificants will enhance the bioavailability of iron; thereby improving the body iron reserves.

A double blind, randomized controlled trail will be conducted on iron deficient female adults (age 18-25 years) in order to determine the synergistic effect of pre-biotics and iron fortificants in anemic human subjects. 75 iron deficient females will be randomly divided into 5 groups (D0, D1, D2, D3 and D4), each having 15 study subjects and will be given varying doses of FeSO4 and NaFeEDTA and Inulin and GOS. Blood samples will be collected from overnight fasted women from each group on monthly basis up to three months. Various biomarkers for iron absorption, LFTs, RFTs, and Immunoglobulins will be estimated.

DETAILED DESCRIPTION:
Study Design A double blind, randomized controlled trial will be used for the purpose of this study.

Study Site The study will be conducted in Islamabad and/or Lahore, depending on the availability of the required sample size with the desired profiles.

Study Duration The trial will last for 12 weeks. Study Population The study population will consist of university going iron deficient female adults (age 18-25 years).

Inclusion and Exclusion Criteria Inclusion Criteria All willing anemic female adults without any chronic diseases such as diabetes or hypertension will be included in the study.

Exclusion Criteria Married females or those with chronic diseases or those already taking iron and/or prebiotic supplements will be excluded from the study.

Sampling Sampling Technique The technique of convenience sampling will be used for the current study. Sample Size Each group will consist of 15 study subjects for the purpose of convenience and the total sample size will be 75.

Treatment Plan For this phase of the study, 4 best treatment combinations of pre-biotics (Inulin & Galactooligosaccharides) and iron fortificants (FeSO4 and NaFeEDTA) will be chosen.

Study participants will be randomly chosen to receive either the best treatment combination 1, 2, 3, 4 or the placebo for 12 weeks on daily basis.

Efficacy Trials Blood samples will be collected from overnight fasted women from each group on monthly basis up to three months. Hematological analysis The collected blood from respective groups will be assessed for hematological analysis.

Iron Biomarkers Obtained sera will also be analyzed for blood serum biomarkers like serum iron, folate, ferritin, transferrin saturation fraction & TIBC.

Liver function tests Liver function tests including AST (Aspartate Aminotransferase), ALT (Alanine Aminotransferase), ALP (Alkaline Phosphatase) and Total Bilirubin will be conducted Renal function tests Blood urea (GLDH-method) and creatinine (Jaffe-method) levels will be determined using commercial kits.

Immunoglobulins Immunoglobulins, including Immunoglobulin A, Immunoglobulin E, Immunoglobulin G, and Immunoglobulin M will be determined using the technique of ELISA (Enzyme linked Immunosorbent Assay).

ELIGIBILITY:
Inclusion Criteria:

* All willing anemic female adults without any chronic diseases such as diabetes or hypertension will be included in the study.

Exclusion Criteria:

* Married females or those with chronic diseases or those already taking iron and/or prebiotic supplements will be excluded from the study.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-04-06 (Actual); Primary Completion 2019-07-06 (Actual); Study Completion 2019-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Waqas Ahmad, PhD, Study Director — University of Veterinary & Animal Sciences, Lahore, Pakistan
Locations (1):
- University of Veterinary and Animal Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
We will see what and how much data will we able to ethically share later on.

RESULTS

PARTICIPANT FLOW:
Groups:
- Prebiotic Inulin & Iron Salt NaFeEDTA: Prebiotic + Iron Forificant: A combination dosage of 963 mg/kg Inulin and 10 ppm NaFeEDTA was given to the study subjects.
- Prebiotic Inulin & Iron Salt NaFeEDTA (2): Prebiotic + Iron Forificant: A combination dosage of 963 mg/kg Inulin and 20 ppm NaFeEDTA was given to the study subjects.
- Prebiotic Inulin & Iron Salt FeS04: Prebiotic + Iron Forificant: A combination dosage of 963 mg/kg Inulin and 30 ppm FeSO4 was given to the study subjects.
- Prebiotic GOS & Iron Salt NaFeEDTA: Prebiotic + Iron Forificant: A combination dosage of 963 mg/kg GOS and 20 ppm NaFeEDTA was given to the study subjects.
Period: Overall Study
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic Inulin & Iron Salt NaFeEDTA (2) | Prebiotic Inulin & Iron Salt FeS04 | Prebiotic GOS & Iron Salt NaFeEDTA
Started | 15 | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic Inulin & Iron Salt NaFeEDTA (2) | Prebiotic Inulin & Iron Salt FeS04 | Prebiotic GOS & Iron Salt NaFeEDTA | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 15 | 15 | 75
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 15 | 15 | 15 | 75
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Pakistan | 15 | 15 | 15 | 15 | 15 | 75

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin Concentration From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
g/dL
  Baseline | 11.44 (0.04) | 11.58 (0.02) | 11.54 (0.01) | 11.61 (0.02) | 11.28 (0.04)
  30 days | 11.52 (0.01) | 11.71 (0.01) | 11.62 (0.01) | 11.78 (0.03) | 11.54 (0.02)
  60 days | 11.64 (0.01) | 11.83 (0.01) | 11.74 (0.01) | 11.90 (0.01) | 11.84 (0.02)
  90 days | 11.91 (0.02) | 12.04 (0.03) | 11.85 (0.01) | 12.17 (0.04) | 12.33 (0.02)

2. Primary Outcome: Change in Hematocrit in Concentration From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: % of RBCs in blood
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
% of RBCs in blood
  Baseline | 30.26 (0.17) | 33.76 (0.19) | 32.77 (0.07) | 33.50 (0.06) | 31.50 (0.06)
  30 days | 31.62 (0.04) | 34.84 (0.12) | 33.72 (0.08) | 34.59 (0.09) | 33.81 (0.13)
  60 days | 32.65 (0.03) | 35.14 (0.10) | 34.76 (0.17) | 35.60 (0.07) | 35.24 (0.06)
  90 days | 34.36 (0.16) | 36.43 (0.07) | 36.17 (0.07) | 36.56 (0.06) | 37.86 (0.26)

3. Primary Outcome: Change in Mean Corpuscular Volume From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
fL
  Baseline | 68.53 (0.11) | 69.56 (0.11) | 73.79 (0.19) | 76.61 (0.13) | 78.06 (0.09)
  30 days | 70.46 (0.29) | 71.63 (0.24) | 74.70 (0.17) | 78.77 (0.14) | 80.03 (0.13)
  60 days | 72.72 (0.09) | 75.11 (0.49) | 80.18 (0.17) | 81.82 (0.17) | 81.96 (0.14)
  90 days | 77.09 (0.15) | 78.64 (0.17) | 83.77 (0.13) | 83.64 (0.15) | 85.59 (0.24)

4. Primary Outcome: Change in Mean Corpuscular Hemoglobin From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
pg
  Baseline | 21.94 (1.35) | 23.63 (1.02) | 20.63 (0.79) | 24.02 (0.69) | 24.56 (0.79)
  30 days | 23.24 (1.14) | 24.83 (0.86) | 21.86 (0.74) | 25.31 (1.08) | 27.42 (0.66)
  60 days | 24.47 (1.00) | 25.05 (0.45) | 24.29 (0.69) | 26.47 (0.28) | 28.26 (0.88)
  90 days | 25.09 (0.89) | 26.76 (0.59) | 26.28 (0.51) | 26.93 (0.26) | 30.75 (0.81)

5. Primary Outcome: Change in Mean Corpuscular Hemoglobin Concentration From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
g/dL
  Baseline | 31.44 (0.77) | 29.30 (0.79) | 28.06 (0.31) | 29.05 (0.50) | 28.51 (0.38)
  30 days | 31.07 (0.74) | 30.30 (1.11) | 30.08 (0.76) | 30.74 (0.67) | 30.67 (0.77)
  60 days | 31.70 (0.45) | 31.91 (0.59) | 31.19 (0.94) | 33.42 (0.96) | 34.25 (0.85)
  90 days | 32.78 (0.58) | 33.46 (0.83) | 33.13 (0.94) | 34.15 (1.06) | 36.91 (0.98)

6. Primary Outcome: Change in Serum Iron Levels From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
mcg/dL
  Baseline | 68.41 (0.70) | 70.97 (0.70) | 72.65 (0.50) | 71.41 (0.60) | 72.60 (0.33)
  30 days | 69.17 (0.85) | 72.34 (1.01) | 73.95 (0.77) | 72.62 (0.73) | 74.51 (0.39)
  60 days | 70.25 (0.85) | 74.34 (1.12) | 75.50 (0.90) | 73.96 (0.99) | 76.61 (0.53)
  90 days | 70.93 (0.95) | 75.36 (1.23) | 77.42 (0.91) | 76.16 (1.09) | 79.10 (0.95)

7. Primary Outcome: Change in Serum Folate Levels From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
ng/mL
  Baseline | 8.74 (0.12) | 9.26 (0.18) | 8.05 (0.08) | 8.96 (0.11) | 8.20 (0.05)
  30 days | 8.81 (0.11) | 10.03 (0.17) | 8.32 (0.10) | 9.40 (0.12) | 9.97 (0.07)
  60 days | 8.88 (0.09) | 10.31 (0.15) | 8.99 (0.11) | 9.75 (0.13) | 10.87 (0.12)
  90 days | 8.94 (0.09) | 10.74 (0.16) | 9.46 (0.13) | 10.02 (0.14) | 11.01 (0.17)

8. Primary Outcome: Change in Serum Ferritin Levels From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
ng/mL
  Baseline | 11.76 (0.11) | 13.73 (0.18) | 13.29 (0.31) | 12.03 (0.09) | 12.67 (0.23)
  30 days | 11.86 (0.08) | 14.09 (0.53) | 13.59 (0.34) | 12.86 (0.10) | 13.56 (0.24)
  60 days | 11.98 (0.09) | 16.28 (0.54) | 14.31 (0.37) | 13.37 (0.14) | 14.77 (0.25)
  90 days | 12.04 (0.17) | 16.88 (0.55) | 15.77 (0.36) | 15.10 (0.27) | 17.55 (0.21)

9. Primary Outcome: Change in Serum Transferrin Levels From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
mg/dL
  Baseline | 16.84 (0.05) | 16.74 (0.09) | 16.38 (0.08) | 16.79 (0.07) | 17.15 (0.06)
  30 days | 16.74 (0.04) | 16.63 (0.09) | 16.30 (0.09) | 16.69 (0.10) | 16.97 (0.04)
  60 days | 16.55 (0.09) | 16.52 (0.11) | 16.21 (0.09) | 16.59 (0.14) | 16.69 (0.16)
  90 days | 16.44 (0.08) | 16.41 (0.13) | 16.09 (0.10) | 16.46 (0.08) | 16.47 (0.12)

10. Primary Outcome: Change in Transferrin Saturation Factor Levels From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: % Transferrin
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
% Transferrin
  Baseline | 16.92 (0.20) | 17.66 (0.24) | 18.49 (0.19) | 17.73 (0.14) | 17.64 (0.10)
  30 days | 17.22 (0.23) | 18.13 (0.32) | 18.91 (0.23) | 18.13 (0.19) | 18.29 (0.13)
  60 days | 17.69 (0.19) | 18.75 (0.38) | 19.41 (0.27) | 18.58 (0.26) | 19.13 (0.16)
  90 days | 17.98 (0.20) | 19.13 (0.42) | 20.05 (0.30) | 19.28 (0.33) | 20.02 (0.27)

11. Primary Outcome: Change in Total Iron Binding Capacity Levels From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
mcg/dL
  Baseline | 404.26 (1.16) | 401.81 (2.12) | 393.06 (1.93) | 402.84 (1.68) | 411.67 (1.53)
  30 days | 401.75 (1.07) | 399.06 (2.19) | 391.08 (2.06) | 400.55 (1.72) | 407.29 (1.61)
  60 days | 397.21 (2.16) | 396.57 (2.62) | 388.93 (2.09) | 398.17 (1.63) | 400.57 (1.52)
  90 days | 394.63 (2.04) | 393.92 (3.17) | 386.16 (2.30) | 395.03 (1.95) | 395.20 (1.75)

12. Secondary Outcome: Change in Liver Functions Tests (ALT) From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
IU/L
  Baseline ALT | 10.51 (0.10) | 11.80 (0.18) | 15.18 (0.44) | 14.73 (0.08) | 11.59 (0.31)
  30 days ALT | 10.61 (0.23) | 11.10 (0.35) | 14.31 (0.52) | 13.24 (0.45) | 10.54 (0.56)
  60 days ALT | 10.59 (0.24) | 10.69 (0.40) | 12.85 (0.76) | 12.32 (0.75) | 9.75 (0.70)
  90 days ALT | 11.28 (0.60) | 10.27 (0.40) | 11.81 (0.84) | 11.13 (0.89) | 9.27 (0.66)

13. Secondary Outcome: Change in Liver Functions Tests (AST) From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
IU/L
  Baseline AST | 16.83 (0.15) | 15.93 (0.53) | 18.07 (0.11) | 18.77 (0.14) | 16.09 (0.26)
  30 days AST | 16.81 (0.14) | 15.76 (0.54) | 17.13 (0.19) | 18.90 (0.82) | 15.99 (0.21)
  60 days AST | 16.68 (0.13) | 15.73 (0.55) | 17.04 (0.22) | 18.80 (0.85) | 15.87 (0.27)
  90 days AST | 16.55 (0.11) | 15.62 (0.56) | 16.84 (0.25) | 18.78 (0.90) | 15.75 (0.32)

14. Secondary Outcome: Change in Liver Functions Tests (ALP) From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
IU/L
  Baseline ALP | 65.84 (1.54) | 69.35 (0.76) | 73.92 (1.33) | 74.99 (1.25) | 68.43 (1.31)
  30 days ALP | 65.63 (2.03) | 71.07 (0.72) | 73.77 (1.32) | 74.86 (1.23) | 68.37 (1.30)
  60 days ALP | 65.51 (1.41) | 73.34 (0.73) | 73.42 (1.36) | 74.72 (1.24) | 68.19 (1.24)
  90 days ALP | 65.48 (1.38) | 76.06 (0.71) | 73.14 (1.35) | 74.55 (1.19) | 68.12 (1.24)

15. Secondary Outcome: Change in Liver Functions Tests (Total Bilirubin) From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
mg/dL
  Baseline Total Bilirubin | 0.31 (0.02) | 0.44 (0.02) | 0.47 (0.02) | 0.61 (0.05) | 0.35 (0.03)
  30 days Total Bilirubin | 0.31 (0.03) | 0.41 (0.03) | 0.43 (0.03) | 0.55 (0.07) | 0.20 (0.04)
  60 days Total Bilirubin | 0.26 (0.04) | 0.36 (0.05) | 0.41 (0.04) | 0.51 (0.08) | 0.13 (0.05)
  90 days Total Bilirubin | 0.19 (0.06) | 0.27 (0.07) | 0.28 (0.07) | 0.43 (0.06) | 0.11 (0.03)

16. Secondary Outcome: Change in Renal Functions Tests (Serum Urea) From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
mg/dL
  Baseline Serum Urea | 18.86 (0.13) | 17.59 (0.19) | 19.60 (0.33) | 21.02 (0.46) | 21.55 (0.27)
  30 days Serum Urea | 18.53 (0.20) | 17.77 (0.18) | 19.63 (0.34) | 21.01 (0.44) | 21.56 (0.29)
  60 days Serum Urea | 18.23 (0.21) | 17.86 (0.17) | 19.65 (0.35) | 21.06 (0.47) | 21.59 (0.31)
  90 days Serum Urea | 18.01 (0.10) | 17.92 (0.20) | 19.10 (2.51) | 21.04 (0.55) | 21.65 (0.35)

17. Secondary Outcome: Change in Renal Functions Tests (Serum Creatinine) From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
mg/dL
  Baseline Serum Creatinine | 0.77 (0.02) | 0.83 (0.02) | 0.89 (0.01) | 0.62 (0.02) | 0.65 (0.02)
  30 days Serum Creatinine | 0.76 (0.03) | 0.86 (0.03) | 0.93 (0.02) | 0.70 (0.04) | 0.74 (0.03)
  60 days Serum Creatinine | 0.78 (0.03) | 0.90 (0.03) | 0.95 (0.02) | 0.77 (0.05) | 0.84 (0.05)
  90 days Serum Creatinine | 0.80 (0.02) | 0.93 (0.03) | 0.92 (0.03) | 0.86 (0.06) | 0.94 (0.03)

18. Secondary Outcome: Change in Immunoglobulins (IgA) From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
g/dL
  Baseline IgA | 200.91 (0.66) | 214.75 (1.39) | 210.56 (1.26) | 204.54 (1.31) | 199.97 (1.34)
  30 days IgA | 201.09 (0.98) | 212.33 (1.82) | 207.42 (2.34) | 201.29 (2.95) | 194.84 (2.56)
  60 days IgA | 198.97 (1.05) | 209.24 (2.06) | 203.48 (4.55) | 198.56 (2.99) | 191.90 (3.65)
  90 days IgA | 196.23 (1.20) | 205.58 (2.75) | 200.37 (4.67) | 195.68 (3.22) | 186.22 (3.65)

19. Secondary Outcome: Change in Immunoglobulins (IgE) From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
IU/mL
  Baseline IgE | 195.02 (1.06) | 184.86 (1.14) | 186.02 (2.81) | 174.62 (1.59) | 193.76 (1.49)
  30 days IgE | 192.59 (1.34) | 181.87 (2.19) | 182.36 (3.44) | 171.73 (2.63) | 189.69 (2.47)
  60 days IgE | 190.81 (1.32) | 179.00 (2.63) | 178.23 (3.79) | 168.62 (3.31) | 185.56 (2.83)
  90 days IgE | 187.32 (1.39) | 176.28 (3.49) | 174.09 (3.50) | 164.60 (3.98) | 177.73 (3.90)

20. Secondary Outcome: Change in Immunoglobulins (IgG) From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
g/dL
  Baseline IgG | 1684.10 (2.39) | 1718.47 (3.49) | 1734.16 (2.61) | 1691.93 (2.76) | 1707.56 (2.14)
  30 days IgG | 1681.23 (2.12) | 1708.98 (5.18) | 1727.20 (3.66) | 1687.67 (3.06) | 1684.95 (2.32)
  60 days IgG | 1678.54 (2.46) | 1704.64 (5.80) | 1719.79 (4.51) | 1682.53 (4.26) | 1655.01 (2.39)
  90 days IgG | 1674.86 (1.86) | 1700.06 (6.47) | 1711.76 (4.32) | 1678.98 (5.66) | 1622.73 (2.45)

21. Secondary Outcome: Change in Immunoglobulins (IgM) From Baseline to 90 Days
Time Frame: Baseline, 30 days, 60 days, 90 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt FeSO4 | Prebiotic GOS & Iron Salt FeSO4 | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic GOS & Iron Salt NaFeEDTA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
g/dL
  Baseline IgM | 303.66 (2.51) | 285.20 (2.57) | 273.74 (2.20) | 267.76 (3.05) | 256.37 (1.69)
  30 days IgM | 300.55 (2.51) | 281.25 (2.36) | 271.15 (2.31) | 264.41 (3.05) | 234.41 (1.87)
  60 days IgM | 299.38 (2.51) | 278.21 (2.59) | 267.81 (2.83) | 259.83 (3.23) | 213.71 (2.28)
  90 days IgM | 296.90 (2.51) | 271.64 (2.93) | 264.02 (3.15) | 256.95 (3.16) | 203.21 (3.43)

ADVERSE EVENTS:
Time Frame: 3 months
Description: The participants were regularly asked if they developed constipation. diarrhea or bloating during the study period, however no one developed such symptoms.
Arm/Group | Placebo Only | Prebiotic Inulin & Iron Salt NaFeEDTA | Prebiotic Inulin & Iron Salt NaFeEDTA (2) | Prebiotic Inulin & Iron Salt FeS04 | Prebiotic GOS & Iron Salt NaFeEDTA
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The research is the property of the University and we have signed an Intellectual Property Rights agreement whereby we will not disclose the study results.

DOCUMENTS (2):
  • Informed Consent Form (2019-01-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT03894449/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT03894449/Prot_SAP_001.pdf